CLINICAL TRIAL: NCT05048927
Title: Symphony IL-6 Cutoff Validation Study for Patients at Risk of Severe Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bluejay Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CES-0003
Record Dates: First submitted 2021-09-09; First posted 2021-09-17 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Severe Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Symphony IL-6 is a device that quantitates human IL-6 by fluorescence enzyme immunoassay (FEIA) from whole-blood specimens. Use of Symphony IL- 6 removes the need for plasma separation before testing. Symphony IL-6 comprises two components, the Symphony Fluorescence Immunoanalyzer and the Symphony IL-6 Cartridge. Whole blood is added to the cartridge and then up to six cartridges can be inserted into the immunoanalyzer. After 20 minutes a readout and printout are given with a quantitative IL-6 concentration. The used cartridges are fully enclosed and can be easily disposed of in general hospital bio-waste. Given the nature of this device and its portability, there is potential for future deployment as a point-of-care (POC) device.

This study is to validate an interleukin-6 (IL-6) cutoff value using the Symphony IL-6 test for patients at high risk of severe sepsis caused by a COVID-19 infection

ELIGIBILITY:
Inclusion Criteria:

* Whole blood specimen collected in EDTA anticoagulant tubes
* Subject is considered to have severe or critical illness per below:

Severe Illness

1. SpO2 < 94% on room air at sea level;
2. Ratio of arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2) < 300 mmHg;
3. Respiratory frequency > 30 breaths/min;
4. Or lung infiltrates >50% Critical Illness

a) Respiratory failure; b) Septic shock; c) And/or multiple organ dysfunction d) At least one criteria of severe illness

* Subject confirmed to be COVID-19 positive by an EUA RT-PCR test
* Subject is 18+ years of age
* Minimum volume of 100µL for Symphony IL-6 testing
* Specimen is available for testing within 12 hours from collection

Exclusion Criteria:

* Subject is receiving an anti-IL-6 treatment
* Subject is receiving corticosteroids
* Hemolyzed specimens

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will test 48 whole blood specimens prospectively collected as baseline samples after admission from confirmed COVID-19 patients at the University of Texas Southwestern Medical Center. Subjects will be symptomatic and have been confirmed by an emergency use authorized (EUA) real-time reverse transcriptase polymerase chain reaction (RT-PCR) test to be COVID-19 positive.
  The whole blood specimens will be de-identified prior to testing on the Symphony IL-6 system. Test results from the Symphony IL-6 system are investigational and are not to be used for managing patient care. The results will not be reported to health care personnel responsible for treating patients.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Validation of IL-6 Cutoff for Patients at High Risk of Severe Sepsis | Specimen is tested within 12 hours from collection
  Validation of the established interleukin-6 concentration in whole blood samples from patients with confirmed COVID-19 infection and are at high risk of severe sepsis

CONTACTS AND LOCATIONS:
Locations (1):
- Tina McCarthy, Acton, Texas, United States